CLINICAL TRIAL: NCT06239428
Title: i-TREAT: An Internet-based Guided Self-help Program for Adolescents and Adults With Other Specified Feeding or Eating Disorders - A Randomized Controlled Trial
Brief Title: i-TREAT: An Internet-based Treatment for Eating Disorders
Acronym: iTREAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region of Southern Denmark (Other)
Collaborators: JaschaFonden (Unknown); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Eik Runge, Principal investigator, Region of Southern Denmark
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 18082179
Record Dates: First submitted 2024-01-19; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Other Specified Feeding or Eating Disorder; Eating Disorder Nos
Keywords: Eating Disorders; Randomized Controlled Trial; Digital intervention; e-Health; Adolescents; Psychiatry
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- i-TREAT (Experimental): The intervention in the experimental group is an internet-based therapist-guided self-help program, called i-TREAT. The program consists of 12 online treatment sessions. It is mainly based on Cognitive Behavior Therapy while inspired by Acceptance and Commitment Therapy. Participants are instructed to complete session-related tasks and receive written feedback from their therapist throughout the treatment. Furthermore, the intervention is also supported by text, illustrations, videos, and a chat function, allowing asynchronous text messaging with the therapist. The treatment courses are expected to run for 12 weeks.
  Interventions: Behavioral: i-TREAT
- Waitlist-control (Active Comparator): Participants randomized to the active waitlist-control group gains access to online mindfulness material for 12 weeks, however, using the material is non-mandatory. After completing the waitlist, participants are offered the i-TREAT intervention. The active waitlist was implemented to prevent potential adverse effects of being on a passive waitlist (which currently comes closest to treatment as usual since no other treatment modalities exist for the target group in the Danish psychiatry).
  Interventions: Other: Waitlist

INTERVENTIONS:
Behavioral: i-TREAT — A 12-session internet-based cognitive behavioral intervention for Danish adolescents and adults with Other Specified Feeding or Eating Disorders.
  Arms: i-TREAT
Other: Waitlist — A 12-week waitlist with access to online mindfulness material.
  Arms: Waitlist-control

SUMMARY:
This clinical study aims to compare the efficacy of an internet-based therapist-guided self-help intervention (named i-TREAT) in reducing eating disorder symptoms in Danish adolescents and adults with Other Specified Feeding or Eating Disorders (OSFED). The study is a randomized controlled trial, comparing the intervention group, receiving i-TREAT, with an active waitlist-control group, receiving online mindfulness material. The investigators hypothesize the intervention group to be superior to the waitlist-control group in terms of 1) reducing eating disorder symptoms and 2) increasing quality of life. The internet-based intervention (i-TREAT) consists of 12 online treatment sessions. It is mainly based on Cognitive Behavior Therapy while inspired by Acceptance and Commitment Therapy. Participants are instructed to complete session-related tasks and receive written feedback from their therapist throughout the treatment.

Furthermore, the intervention is also supported by text, illustrations, videos, and a chat function, allowing asynchronous text messaging with the therapist. The treatment courses are expected to run for up to 12 weeks. Participants completing the 12-week waitlist are subsequently offered the i-TREAT intervention. The investigators expect to include 63 participants in each group, who will be recruited through 1) self-referral on the project's website and 2) referral from mental health institutions and doctors.

DETAILED DESCRIPTION:
1. Intervention (i-TREAT)

   The online treatment program (i-TREAT) consists of 12 sessions developed in cooperation with clinical psychologists and technical staff and is hosted on the digital platform MindDistrict that can be accessed by computer or mobile app. The text-based treatment content is supported by videos and illustrations, which is recommended by Andersson. The treatment is based on cognitive behavioral therapy that has been widely used in other international eating disorder treatments. Thus, the treatment sessions include psychoeducation about eating disorders, treatment-related tasks, such as observation of their behavior in real time and identifying perpetuating and maintaining factors, establishing coping strategies and behavioral changes, and receiving written support from a clinician.

   Patients will be guided through the treatment by a clinician specialized in eating disorders. Clinicians are providing written feedback for the patient after completion of each session. The feedback must be sent no later than seven days after session completion. Additionally, patients can communicate with their therapist though an asynchronous chat function, supported by a feature enabling the patients to invite relatives to the chat as well. This feature is vital, as adolescents will be required to involve their parents in the treatment process. However, unlike family therapy, which actively involves the parents to take responsibility for the treatment and control of their child's eating, Enhanced Cognitive Behavioral Therapy (CBT-E) for adolescents with eating disorders gives more autonomy to the patient and changes the parents' role to being more supportive rather than directive. This is one of the features of internet-based Cognitive Behavioral Therapy (iCBT), which makes it suitable for younger patients, as it fits their needs and concerns about control, while promoting independence and autonomy. The internet-based treatment format further strengthens these benefits. In the asynchronous chat function, patients can discuss with the therapist and parents how the parents may assist the patient in establishing changes while informing the parents about the treatment and child's progress. Furthermore, patients may address questions or comments about treatment content or tasks, personal experiences, motivational issues etc. It is also possible to permanently save all content and tasks on their hardware.

   The treatment program is both available on web-browser and app.
2. Methods

2.1. Design

The study is a randomized controlled trial consisting of two conditions:

1. Experimental group receiving i-TREAT over 12 weeks.
2. Active waitlist-control group receiving online mindfulness exercises for 12 weeks.

   Participants randomized to the control group will be offered i-TREAT after completing the waitlist. Thus, the randomized controlled trial follows a delayed cross-over design (also called waitlist control design).

   2.2. Randomization

   An independent datamanager from the Open Patient data Explorative Network, Department of Clinical Medicine, University of Southern Denmark (OPEN), who is not involved in the trial, will perform the randomization. A computerized random number generator will be used to generate a random allocation sequence. A computerized random number generator will be applied with an allocation ratio of 1:1. Participants will be stratified by age in two categories: 15-17 years of age and ≥ 18 years of age respectively. Block randomization will be used with variable block sizes. The allocation sequence will be blinded for all involved researchers until the point of interpreting the results.

   2.3. Time frame

   The trial phase will commence in the beginning of September 2024 and close in the end of February 2026 (last patient last visit). A typical treatment course will run for approximately 12 weeks, as one session intentionally takes one week to complete. However, the overall time may deviate from this estimation, as clinicians also use time for writing feedback and some patients may be require or feel a need to repeat a given session (or sessions). After treatment completion, patients will still have access to the treatment program at least three months afterwards, where they are invited to complete follow-up questionnaires but they will not be able to correspond with their therapist during this period.

   Data analysis will take place between January 2026 and October 2026. If the project yields positive results, a process will be started on implementing the treatment as part of the clinic at the Centre for Digital Psychiatry.
3. Statistics

   The estimated sample size was calculated based on an expected mean difference score of 0.8 on the Eating Disorder Examination Questionnaire (EDE-Q) global score (primary measure score) in the intervention group. The expected score was based on results of EDE-Q global mean difference scores from other studies delivering iCBT for OSFED: ter Huurne et al. with a score of 0.7; Strandskov et al. with a score of 0.79; and Ruwaard et al. with a score of 1.5. Power analysis revealed a sample size of 50 participants in each group based on significance level of 5% and a power of 80%. Taking 20% drop-out rates into account, the investigators aim to invite 63 participants in each group.

   Statistical analyses will be carried out using SPSS version 21. Chi square or Fisher's exact tests will be used to compare categorical measures between the groups, and t-tests or Mann-Whitney tests will be used to compare continuous measures. In terms of determining the efficacy of the intervention, Mixed Models for repeated measures will be used, based on statistical comparisons between the pre-treatment and post-treatment EDE-Q score of the patients included in treatment and compared to the active control group.

   Between-group effect sizes will be calculated using Cohen's d.
4. Recruitment

The investigators aim to recruit participants from specific risk groups:

1. Participants (from the whole country) with eating disorder symptoms, seeking online treatment as a first step.
2. Patients with OSFED rejected from the mental health hospitals or patients recovering from eating disorders in the Region of Southern Denmark (eating disorder units for children/adolescents and adults in Odense and Vejle).

Recruitment will be done in collaboration with patient organizations (Foreningen Spiseforstyrrelser og Selvskade and Askovhus) and through advertisement on the website and social media of the Centre for Digital Psychiatry. Participants can apply for treatment from the website at Centre for Digital Psychiatry and do not need a referral from their medical doctor. The application form consists of an online survey with eating disorder assessment and quality of life measures. The EDE-Q will be the primary assessment tool. The questionnaire is based on the Eating Disorder Examination Interview (EDE-I), which is the gold standard instrument to assess symptoms of eating disorders. The two clinicians will evaluate the submitted electronically forms and decide for preliminary inclusion.

Participants eligible for treatment will be contacted by telephone by a member of the research team and informed about the study and provided with a written consent form if interested. The participants will be notified that they have the right to reflecting time, and that they can turn in the consent form with in one week from the phone call. If the participants turn in the consent form within a week, a member of the research team will call them back to get the oral consent. The phone call will be made in CEDIP's facilities where it can be completed undisturbed. For participants between the ages of 15 to 17 years, written information about the project will also be sent to the parents and they will also need to participate in the telephone screening. If the participant comes of age (18 years old) during the trial, independent consent will be obtained. They will be informed that they can withdraw at any time from the treatment and/or the study without any need of explanation and without consequences for other normal treatment options. If the participant is excluded after the final screening, they will be asked for consent on us using their data from the screening. This will be done due to the importance of knowing why participants are excluded from the trial. Participants will not receive any financial compensation for their participation in the study. Finally, they will be randomly assigned to the intervention group or the control group, and commence treatment.

Participants will not receive any financial compensation for participating in the study.

5. Risks, side effects and safety procedure

There are no known risks or negative side effects of the digital program. However, the patient group is considered vulnerable, and the program content may be challenging and cause fluctuations in symptoms. Thus, it is most important to mention that the participants will be monitored by the research team (intervention and waitlist control group) and the affiliated psychologist (intervention group only). Furthermore, participants will be introduced to an emergency contact list at the very first session in the program. The investigators will also inform the participants about these risks and make sure they are familiar with the study frame.

6. The processing of personal information

Any personally sensitive information is processed by Centre for Digital Psychiatry in personally identifiable form for as long as it is necessary for the research purpose. The storages of information are in accordance with responsible research practice and in relation to general data protection regulation. When the information is no longer necessary for the research project, it will be anonymized.

7. Funding

Centre for Digital Psychiatry, represented by the director, Mrs. Marie Paldam Folker, has taken initiative to the project. The principal investigator, Eik Runge, has been responsible for fund raising and conducting applications for project approvals.

The project is funded by five different sponsors: JaschaFonden (350.000kr.); Psykiatriens Forskningsfond (562.500kr.); PhD scholarship from the University of Southern Denmark (512.500kr.); PhD scholarship from the Mental Health Services in the Region of Southern Denmark (612.500kr.); and a deficit guarantee from the Centre for Digital Psychiatry (868.700kr.).

Most of the funds (2.500.000kr.) are used on salaries to the PhD student (full time) and two clinicians (part time) running the treatment. The remaining amount is used on other costs, such as software maintenance, program licenses, and tuition and publication fees. The funds are administrated partially at the University of Southern Denmark, Faculty of Health Sciences (only salary for the PhD student the first year) and the Psychiatry in the Region of Southern Denmark, Centre for Digital Psychiatry (rest of the funds, including salary and other costs for the last two years).

The PhD student and principal investigator, Eik Runge, has no economic affiliations to the sponsors or other stakeholders.

8. Dissemination plan

After the trial and evaluation, the investigators will conduct a report, including all results of the project. The report will be made publicly available on the website of Centre for Digital Psychiatry and the Mental Health Services in the Region of Southern Denmark. Furthermore, as part of a PhD program, three scientific papers will be produced and published, utilizing data from the project. Lastly, the results will be orally and visually presented at various national as well as international conferences. All data will be anonymized across reports, papers, and presentations.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 15 to 17 years, or age ≥ 18 years.
2. Fulfilment of the diagnostic criteria for Other Specified Feeding or Eating Disorders according to DSM-V and ICD-11.
3. Comprehension of the Danish language.
4. Consent from at least one parent for participants between 15 to 17 years.
5. Access to the Danish secure mail system E-boks.

Exclusion Criteria:

1. Body Mass Index (BMI) ≤ 17,5.
2. Lack of access to technological device (computer and tablet/iphone/android).
3. Concurrent participation in other psychotherapeutic treatment.
4. Concurrent diagnosis of severe depression, severe anxiety, or substance dependence disorder.
5. Previously diagnosed with psychosis or Autism Spectrum Disorder.
6. If on medication, medication must be stable for six months prior to, as well as during, the study participation (i.e., no changes in type of medication or dosage).

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Eating Disorder Examination Questionnaire (EDE-Q) | Baseline (Day 0), mid-treatment (up to six weeks), post-treatment (up to 12 weeks), and follow-up (three months)
  The Eating Disorder Examination Questionnaire (EDE-Q) is a self-report questionnaire assessing the severity and type of eating disorder symptoms and psychopathology during the preceding 28 days. The current version is designed to generate Diagnostic and Statistical Manual of Mental Disorders (DSM-5) compatible eating disorder diagnoses. Finally, the EDE-Q has an excellent internal consistency reliability (Cronbach's α = .95) and is considered the gold standard for measuring eating disorder psychopathology.

SECONDARY OUTCOMES:
SCOFF Questionnaire | Baseline (Day 0), mid-treatment (up to six weeks), post-treatment (up to 12 weeks), and follow-up (three months)
  The SCOFF Questionnaire is a 5-item scale used to screen for eating disorder symptoms, and the name is an acronym for the keywords in each item (Sick, Control, One stone, Fat, Food). The SCOFF has shown good validity and reliability in both adults and adolescents. It has also been translated and validated in a Danish version.
Major Depression Inventory (MDI) | Baseline (Day 0), mid-treatment (up to six weeks), post-treatment (up to 12 weeks), and follow-up (three months)
  The Major Depression Inventory (MDI) is a 10-item questionnaire pertaining to the International Classification of Diseases (ICD-10) and DSM-5 symptoms of depression illness. For each of the three final items (items 8-10), the item is divided into two sub-items, of which only the sub-item with the highest score is included. The scale measures items on a 6-point scale from 0 (never) to 5 (all the time) over the last two weeks. The MDI global score ranges from 0 (no symptoms of depression) to 50 (extreme symptoms of depression) and describes the severity of depressive symptoms present in the patient.
EuroQol - 5 Dimension - 5 Level (EQ-5D-5L) | Baseline (Day 0), mid-treatment (up to six weeks), post-treatment (up to 12 weeks), and follow-up (three months)
  Quality of life is measured with the EuroQol - 5 Dimension - 5 Level (EQ-5D-5L). The EQ-5D-5L is a self-report questionnaire comprised of five items, answered on a scale from 0 (no problems) to 4 (severe problems). The items cover five domains: mobility, selfcare, usual activities, pain/discomfort, and anxiety and depression. In addition to the five items, respondents will answer a visual analogue scale (VAS), ranging from 0 (worst imaginable health) to 100 (best imaginable health).

OTHER OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Baseline (Day 0), session 1, session 2, session 3, session 4, session 5, mid-treatment (up to six weeks), session 7, session 8, session 9, session 10, session 11, post-treatment (up to 12 weeks), and follow-up (three months)
  Depression and suicide risk is measured with the Patient Health Questionnaire (PHQ-9). The PHQ-9 is a self-report questionnaire comprised of nine items, answered on a 4-point Likert scale from 0 (not at all) to 3 (nearly every day). The PHQ-9 shows good psychometric properties. The last item of the scale addresses passive suicide risk, which is the main reason why this questionnaire was included.
Credibility/Expectancy Questionnaire | Baseline (Day 0), session 1, session 3, mid-treatment (up to six weeks), session 9
  The Credibility/Expectancy Questionnaire is used to assess the participants' credibility and expectations related to the treatment. The scale consists of 6 items divided into two subscales; one consisting of four "think" questions and one consisting of two "feel" questions. The scale has been validated across different populations with Cronbach's α ranging from 0.79 and 0.93 and a test-retest reliability (r) ranging from 0.75 to 0.82.
Compliance | Session 1, session 2, session 3, session 4, session 5, mid-treatment (up to six weeks), session 7, session 8, session 9, session 10, session 11, post-treatment (up to 12 weeks)
  Compliance will be assessed by the therapists, rating the quantity compliance (the percentage of assigned treatment tasks completed: 0-100%) and quality compliance (overall quality of treatment task performance on a Likert scale from 0-5) at each session. A study by Schmidt & Woolaway-Bickel has proven therapist ratings of compliance to be superior to patient ratings in terms of predicting symptom reduction.
Adherence | Post-treatment (up to 12 weeks) or at drop-out (any time point between Day 0 and up to 12 weeks)
  Adherence will be assessed by reporting the percentage of sessions completed by the patient. Patients will be considered completers when completing all 12 sessions and fulfilling the post-treatment questionnaires. Drop-outs will be categorized into early treatment drop-outs (before session 6) and late treatment drop-outs (after session 6).
Client Satisfaction Questionnaire (CSQ-8) | Post-treatment (up to 12 weeks)
  General satisfaction with the received treatment will be measured with the Client Satisfaction Questionnaire - 8 (CSQ-8). The CSQ-8 consists of 8 items, answered on a scale from 1 to 4.
Negative Effects Questionnaire (NEQ) | Post-treatment (up to 12 weeks)
  Potential adverse effects or symptoms of deterioration is measured with the Negative Effects Questionnaire (NEQ). The scale consists of 32 items and has shown acceptable psychometric properties.
System Usability Scale (SUS) | Post-treatment (up to 12 weeks)
  Accessibility and user-friendliness of the online program will be measured with the System Usability Scale (SUS). The SUS is a 10-item self-report scale, probing the user's experiences with a given system. Items are answered on a scale from 1 (strongly disagree) to 5 (strongly agree), with a total score range from 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Marie P Folker, Cand.scient., Study Chair — Centre for Digital Psychiatry
Locations (1):
- Centre for Digital Psychiatry, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data that underlie results in the study-related articles will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available once the study ends ultimo 2026.
Access Criteria: The data can be accessed through open access supplementary material or upon request from the corresponding author(s).

REFERENCES:
- [Background] Fairburn CG, Beglin SJ. Assessment of eating disorders: interview or self-report questionnaire? Int J Eat Disord. 1994 Dec;16(4):363-70. PMID 7866415
- [Background] Fairburn, C. G. (2008). Cognitive Behavior Therapy and Eating Disorders. Guilford Press.
- [Background] World Health Organization (1992). The ICD-10 Classification of Mental and Behavioural Disorders. Clinical descriptions and diagnostic guidelines. World Health Organization.
- [Background] Aardoom JJ, Dingemans AE, Slof Op't Landt MC, Van Furth EF. Norms and discriminative validity of the Eating Disorder Examination Questionnaire (EDE-Q). Eat Behav. 2012 Dec;13(4):305-9. doi: 10.1016/j.eatbeh.2012.09.002. Epub 2012 Sep 19. PMID 23121779
- [Background] Botella J, Sepulveda AR, Huang H, Gambara H. A meta-analysis of the diagnostic accuracy of the SCOFF. Span J Psychol. 2013;16:E92. doi: 10.1017/sjp.2013.92. PMID 24230955
- [Background] Lichtenstein MB, Hemmingsen SD, Stoving RK. Identification of eating disorder symptoms in Danish adolescents with the SCOFF questionnaire. Nord J Psychiatry. 2017 Jul;71(5):340-347. doi: 10.1080/08039488.2017.1300322. Epub 2017 Mar 14. PMID 28290749
- [Background] Bech, P. (2012). Clinical Psychometrics. John Wiley & Sons, Ltd.
- [Background] Feng YS, Kohlmann T, Janssen MF, Buchholz I. Psychometric properties of the EQ-5D-5L: a systematic review of the literature. Qual Life Res. 2021 Mar;30(3):647-673. doi: 10.1007/s11136-020-02688-y. Epub 2020 Dec 7. PMID 33284428
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Nielsen, M. D., Andreasen, C., & Thastum, M. (2016). A Danish study of One-session Treatment for Specific Phobias in Children and Adolescents. Scandinavian Journal of Child and Adolescent Psychiatry and Psychology, 4, 65-76. https://doi.org/10.21307/sjcapp-2016-011
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Schmidt NB, Woolaway-Bickel K. The effects of treatment compliance on outcome in cognitive-behavioral therapy for panic disorder: quality versus quantity. J Consult Clin Psychol. 2000 Feb;68(1):13-8. doi: 10.1037//0022-006x.68.1.13. PMID 10710836
- [Background] Rozental A, Kottorp A, Forsstrom D, Mansson K, Boettcher J, Andersson G, Furmark T, Carlbring P. The Negative Effects Questionnaire: psychometric properties of an instrument for assessing negative effects in psychological treatments. Behav Cogn Psychother. 2019 Sep;47(5):559-572. doi: 10.1017/S1352465819000018. Epub 2019 Mar 15. PMID 30871650
- [Background] Brooke, J. (1996). SUS: A
- [Background] Atwood ME, Friedman A. A systematic review of enhanced cognitive behavioral therapy (CBT-E) for eating disorders. Int J Eat Disord. 2020 Mar;53(3):311-330. doi: 10.1002/eat.23206. Epub 2019 Dec 16. PMID 31840285
- [Background] ter Huurne ED, Postel MG, de Haan HA, DeJong CA. Effectiveness of a web-based treatment program using intensive therapeutic support for female patients with bulimia nervosa, binge eating disorder and eating disorders not otherwise specified: study protocol of a randomized controlled trial. BMC Psychiatry. 2013 Nov 16;13:310. doi: 10.1186/1471-244X-13-310. PMID 24238630
- [Background] Andersson G. Internet-Delivered Psychological Treatments. Annu Rev Clin Psychol. 2016;12:157-79. doi: 10.1146/annurev-clinpsy-021815-093006. Epub 2015 Dec 11. PMID 26652054
- [Background] Ter Huurne ED, de Haan HA, Postel MG, DeJong CAJ, VanDerNagel JEL, van der Palen J. Long-term effectiveness of web-based cognitive behavioral therapy for patients with eating disorders. Eat Weight Disord. 2021 Apr;26(3):911-919. doi: 10.1007/s40519-020-00929-0. Epub 2020 May 24. PMID 32449152
- [Background] Strandskov SW, Ghaderi A, Andersson H, Parmskog N, Hjort E, Warn AS, Jannert M, Andersson G. Effects of Tailored and ACT-Influenced Internet-Based CBT for Eating Disorders and the Relation Between Knowledge Acquisition and Outcome: A Randomized Controlled Trial. Behav Ther. 2017 Sep;48(5):624-637. doi: 10.1016/j.beth.2017.02.002. Epub 2017 Mar 2. PMID 28711113
- [Background] Ruwaard J, Lange A, Broeksteeg J, Renteria-Agirre A, Schrieken B, Dolan CV, Emmelkamp P. Online cognitive-behavioural treatment of bulimic symptoms: a randomized controlled trial. Clin Psychol Psychother. 2013 Jul-Aug;20(4):308-18. doi: 10.1002/cpp.1767. Epub 2012 Feb 1. PMID 22298417